CLINICAL TRIAL: NCT01201967
Title: A Collaborative Care Program to Improve Treatment of Depression and Anxiety Disorders in Cardiac Patients (MOSAIC)
Brief Title: A Collaborative Care Program to Improve Treatment of Depression and Anxiety Disorders in Cardiac Patients
Acronym: MOSAIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director, Blake 11, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010P-001414
Record Dates: First submitted 2010-09-07; First posted 2010-09-15 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Depression; Generalized Anxiety Disorder; Panic Disorder
Keywords: Collaborative care; Cardiovascular disease; Depression; Anxiety
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder; Panic Disorder; Cardiovascular Diseases; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative care (Experimental): Study care manager provides education and coordinates treatment between study psychiatrist, patient, and primary medical physician. This occurs in the hospital and by phone after discharge. Care manager may also provide phone-based therapy.
  Interventions: Other: Collaborative care
- Usual care (Placebo Comparator): Patient's physicians are informed of diagnosis of depression/anxiety disorder
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Collaborative care — Study care manager provides psychoeducation, therapy, and care coordination between patient, psychiatrist, and primary medical physicians.
  Arms: Collaborative care
Other: Usual care — Patient's primary medical physician informed of mental health symptoms/diagnosis
  Arms: Usual care

SUMMARY:
For this trial, the investigators propose a prospective trial of a collaborative care program to identify and treat depression, generalized anxiety disorder, and panic disorder among patients admitted to the hospital for an acute cardiac illness (acute coronary syndrome, congestive heart failure, or arrhythmia). Such assessment and treatment for depression/generalized anxiety disorder/panic disorder will begin in the hospital, and ongoing management will continue for six months following discharge.

The investigators hypothesize that this model will lead to increased treatment rates, improved mood, reduced anxiety, and improved medical outcomes in this vulnerable population. If this model is effective, it could be implemented clinically to provide better and more complete care to patients hospitalized with acute cardiac illness, for whom depression and anxiety may be a risk factor for complications and death.

This will be a two-arm, single-blind randomized controlled trial, with one-half of patients randomized to collaborative care and one-half randomized to the control condition (usual care). Psychiatric treatment in the intervention arm will be provided in concert with patients' primary care physicians-with primary care physicians prescribing all medications-within a framework supervised by a psychiatrist.

The investigators will enroll patients who have any (or all) of the three included psychiatric diagnoses to improve the utility of the intervention. The investigators have chosen to enroll patients with several different cardiac diagnoses. This will allow the researchers to include patients with heterogeneous diagnoses and illness severity to determine if our intervention is effective in a broad population of patients with heart disease. The investigators will study an intervention targeting depression, generalized anxiety disorder, and panic disorder: all three disorders are disabling and associated with adverse cardiovascular outcomes, treatments for the conditions are highly similar, the investigators can treat patients who have more than one disorder, and a prior outpatient program successfully simultaneously addressed more than one mental health condition.

The project will involve: (1) screening patients for depression, generalized anxiety disorder, and panic disorder as part of usual clinical care, (2) evaluation of positive-screen patients by a study social work care manager, (3) a multicomponent in-hospital intervention (for collaborative care patients) that involves patient education, specialist-provided treatment recommendations, and a goal of in-hospital treatment initiation, and (4), after discharge, continued phone-based evaluation and care coordination with primary care physicians to provide stepwise treatment in the collaborative care arm. The intervention has been designed to be low-cost, low-burden, and easily generalizable to other settings.

DETAILED DESCRIPTION:
* Primary in-hospital outcome measure:

  - Adequate treatment by discharge (percent rates)
* Primary overall study measure:

  - Change from baseline mental health-related quality of life (Short Form-12 Mental Component Score)
* Depression outcome measures:

  - Change from baseline depression (Patient Health Questionnaire-9)
* Anxiety outcome measures:

  - Change from baseline anxiety (Hospital Anxiety and Depression Scale-Anxiety Subscale)
* Medical outcome measures:

  * Change from baseline physical function (Duke Activity Status Index)
  * Change from baseline adherence (Medical Outcomes Study Specific Adherence Scale)
  * Change from baseline physical health-related quality of life (Short Form-12 Physical Component Score)
  * Change in rates of cardiac rehospitalizations at 24 weeks (exploratory aim)

    * 24 weeks is primary endpoint for all post-discharge analyses *

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18-up)admitted to inpatient cardiac unit at Massachusetts General Hospital
* Primary diagnosis of acute coronary syndrome, congestive heart failure, or arrhythmia
* Positive anxiety or depression screen during initial nursing intake interview that is performed as part of usual clinical care
* Meets criteria for clinical depression, generalized anxiety disorder, or panic disorder

Exclusion Criteria:

* Bipolar disorder
* Substance use disorder
* Psychosis
* Cognitive disorder
* Active suicidal ideation
* Medical condition with likely survival less than 6 months
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Huffman JC, Mastromauro CA, Beach SR, Celano CM, DuBois CM, Healy BC, Suarez L, Rollman BL, Januzzi JL. Collaborative care for depression and anxiety disorders in patients with recent cardiac events: the Management of Sadness and Anxiety in Cardiology (MOSAIC) randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):927-35. doi: 10.1001/jamainternmed.2014.739. PMID 24733277
- [Derived] Celano CM, Suarez L, Mastromauro C, Januzzi JL, Huffman JC. Feasibility and utility of screening for depression and anxiety disorders in patients with cardiovascular disease. Circ Cardiovasc Qual Outcomes. 2013 Jul;6(4):498-504. doi: 10.1161/CIRCOUTCOMES.111.000049. Epub 2013 Jun 11. PMID 23759474

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Collaborative Care | Usual Care
Started | 92 | 91
Completed | 86 | 86
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis was employed. All randomized participants were included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Collaborative Care | Usual Care | Total
Number analyzed (Participants) | 92 | 91 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (12.7) | 60.1 (12.8) | 60.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 49 | 48 | 97
Region of Enrollment [Number; unit: participants]
  United States | 92 | 91 | 183
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 is a 9-item scale that measures depression severity. Each question asks how often the subject experiences symptoms of depression and offers four answers: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. Scores are totaled and range from 0-27. To be considered depressed, subjects had to (a) have a total score of 10 or more, (b) answer five questions with a score of 2 or 3, and (c) one of the five questions had to be question 1 or question 2 (or both). Anyone who did not meet these criteria were not considered depressed.
  units on a scale | 15.9 (4.2) | 15.6 (5.0) | 15.8 (4.6)
Hospital Anxiety and Depression Scale - Anxiety Subscale [Mean (Standard Deviation); unit: units on a scale] — The HADS-A is a 7-item scale used to measure anxiety severity. Each question asks about a specific symptom of anxiety and offers four answers: 0 = Never / Not at all, 1 = A little / Time to time, 2 = Quite often / Usually, 3 = Most of the time / Very often. Scores are totaled and range from 0-21. A higher score means more anxiety.
  units on a scale | 10.9 (4.0) | 11.5 (3.9) | 11.2 (3.9)
Duke Activity Status Index [Mean (Standard Deviation); unit: units on a scale] — The DASI is a 12-item scale that measures physical function. Each question asks about whether the subject can complete a physical activity and are given the following options: Scores range from 0 to 58.2. Lower scores indicate lower levels of physical function.
  units on a scale | 19.7 (15.8) | 21.4 (16.9) | 20.5 (16.3)
Medical Outcomes Study - Specific Adherence Scale [Mean (Standard Deviation); unit: units on a scale] — The MOS-SAS is a 3-item scale used to assess medication adherence, physical activity adherence, and diet adherence. Each question asks how often the subject adheres to the behavior, providing the following options: 1 = None of the time, 2 = A little of the time, 3 = Some of the time, 4 = A good bit of the time, 5 = Most of the time, 6 = All of the time. Scores are totaled and range from (3 to 18). A low score indicates poorer adherence to healthy behaviors.
  units on a scale | 13.0 (3.5) | 14.2 (3.1) | 13.6 (3.3)
SF-12 Mental Component Score [Mean (Standard Deviation); unit: units on a scale] — The SF-12 Mental Component Score is a 6-item scale that assesses mental health-related quality of life. Each question provides the option of 2-6 answers. Some questions are Yes/No (2 options), while others ask how often something occurs (6 options, etc.). Scores are calculated using a formula and can range from 0 to 100. A score of 50 indicates average mental health-related quality of life. Higher scores represent higher than average mental health-related quality of life, and lower scores represent lower mental health-related quality of life.
  units on a scale | 34.2 (9.7) | 36.3 (8.9) | 35.2 (9.3)
SF-12 Physical Component Score [Mean (Standard Deviation); unit: units on a scale] — The SF-12 Physical Component Score is a 6-item scale that assesses physical health-related quality of life. Each question provides the option of 2-6 answers. Some questions are Yes/No (2 options), while others ask how often something occurs (6 options, etc.). Scores are calculated using a formula and can range from 0 to 100. A score of 50 indicates average physical health-related quality of life. Higher scores represent higher than average physical health-related quality of life, and lower scores represent lower physical health-related quality of life.
  units on a scale | 32.9 (10.8) | 33.8 (11.0) | 32.9 (10.5)
Euro Quality of Life-5 Domain [Mean (Standard Deviation); unit: units on a scale] — The Euro Quality of Life-5 Domain is a 5-item scale that assesses quality of life. Each question asks about difficulties with certain areas of health (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and offer three possible answers: No problems, Moderate problems, Extreme problems. Scores can range from 0.000-1.000, with lower scores indicating less quality of life, and higher scores indicating higher quality of life.
  units on a scale | 0.40 (0.34) | 0.44 (0.33) | 0.42 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mental Health-related Quality of Life From Baseline to 24 Weeks
Description: Mental health-related quality of life is measured by the Short Form-12 Mental Component Score (SF-12 MCS). The SF-12 MCS is a 6-item scale that assesses mental health-related quality of life. Each question provides the option of 2-6 answers. Some questions are Yes/No (2 options), while others ask how often something occurs (6 options, etc.). Scores are calculated using a formula and can range from 0 to 100. A score of 50 indicates average mental health-related quality of life. Higher scores represent higher than average mental health-related quality of life, and lower scores represent lower mental health-related quality of life.
Time Frame: Baseline, 24 weeks
Population: 92 participants in the Collaborative Care group were compared to 91 participants in the Usual Care group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
units on a scale | 8.87 [5.67 to 12.06] | 8.39 [5.38 to 11.40]
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 5.68, 95% CI 2-sided [2.14 to 9.22]

2. Secondary Outcome: Change in Depression Symptoms From Baseline to 24 Weeks
Description: Depression symptoms measured by the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item scale that measures depression severity. Each question asks how often the subject experiences symptoms of depression and offers four answers: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. Scores are totaled and range from 0-27. To be considered depressed, subjects had to (a) have a total score of 10 or more, (b) answer five questions with a score of 2 or 3, and (c) one of the five questions had to be question 1 or question 2 (or both). Anyone who did not meet these criteria were not considered depressed.
Time Frame: Baseline, 24 weeks
Population: 92 participants in the Collaborative Care group were compared to 91 participants in the Usual Care group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
units on a scale | -6.99 [-8.61 to -5.36] | -7.67 [-9.04 to -6.30]
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis; Mean Difference (Final Values) = -2.05, 95% CI 2-sided [-4.06 to -0.05]

3. Secondary Outcome: Change in Anxiety Symptoms From Baseline to 24 Weeks
Description: Anxiety symptoms measured with the Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A). The HADS-A is a 7-item scale used to measure anxiety severity. Each question asks about a specific symptom of anxiety and offers four answers: 0 = Never / Not at all, 1 = A little / Time to time, 2 = Quite often / Usually, 3 = Most of the time / Very often. Scores are totaled and range from 0-21. A higher score means more anxiety.
Time Frame: Baseline, 24 weeks
Population: 92 participants in the Collaborative Care group were compared to 91 participants in the Usual Care group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
units on a scale | -3.43 [-4.62 to -2.24] | -4.85 [-5.94 to -3.76]
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.93 to 1.76]

4. Secondary Outcome: Rate of Adequate Treatment of Depression and/or Anxiety Symptoms 5 Days After Enrollment
Description: Adequate treatment was defined as:
  (1) Prescription of a standard dose of an established first-line treatment for depression, generalized anxiety disorder, or panic disorder, and/or (2) referral to evidence-based psychotherapy (either to an outside mental health provider or a Cognitive Behavioral Therapy workbook in the Collaborative Care arm of the study).
  Patients already engaged in #1 and/or #2 at the time of enrollment had a different process. Subjects must have been engaged in at least 4 weeks of treatment prior to enrollment while still meeting criteria for the disorder. For this population, adequate treatment was defined as:
  (1) Prescription dose increase/augmentation/switch, and/or (2) referral to psychotherapy (either to an outside mental health provider or a Cognitive Behavioral Therapy workbook in the Collaborate Care arm).
  Timeframe of "5 days after enrollment" was determined by calculating the median length of hospitalization for all subjects.
Time Frame: 5 days after enrollment
Population: 92 participants in the Collaborative Care group were compared to 91 participants in the Usual Care group.
Measure: Number; unit: participants
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
participants | 69 | 6
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Ratio (RR) = 11.4, 95% CI 2-sided [5.20 to 24.9]

5. Secondary Outcome: Change in Adherence to Health Behaviors From Baseline to 24 Weeks
Description: Adherence to health behaviors is measured with the Medical Outcome Study Specific Adherence Scale (MOS-SAS). The MOS-SAS is a 3-item scale used to assess medication adherence, physical activity adherence, and diet adherence. Each question asks how often the subject adheres to the behavior, providing the following options: 1 = None of the time, 2 = A little of the time, 3 = Some of the time, 4 = A good bit of the time, 5 = Most of the time, 6 = All of the time. Scores are totaled and range from (3 to 18). A low score indicates poorer adherence to healthy behaviors.
Time Frame: Baseline, 24 weeks
Population: 92 participants in the Collaborative Care group were compared to 91 participants in the Usual Care group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
units on a scale | 2.2 [1.30 to 3.10] | 1.70 [0.80 to 2.59]
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.28, Mixed Models Analysis; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.51 to 1.76]

6. Secondary Outcome: Number of Rehospitalizations From Baseline to 24 Weeks
Description: The number of rehospitalizations from baseline to 24 weeks was measured by contacting subjects' medical providers at 24 weeks and by asking subjects about rehospitalizations during each follow-up phone call.
Time Frame: 24 weeks
Measure: Number; unit: readmissions
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
readmissions | 29 | 30
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.83, Chi-squared; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.63 to 1.46]

7. Secondary Outcome: Change in Health Status From Baseline to 24 Weeks
Description: Health status measured by the Euro Quality of Life-5 Domain (EQ5D). The EQ5D is a 5-item scale that assesses quality of life. Each question asks about difficulties with certain areas of health (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and offer three possible answers: No problems, Moderate problems, Extreme problems. Scores can range from 0.000-1.000, with lower scores indicating less quality of life, and higher scores indicating higher quality of life.
Time Frame: Baseline, 24 weeks
Population: 92 participants in the Collaborative Care group were compared to 91 participants in the Usual Care group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
units on a scale | 0.16 [0.08 to 0.23] | 0.18 [0.10 to 0.27]
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.012 to 0.22]

8. Secondary Outcome: Change in Physical Function From Baseline to 24 Weeks
Description: Physical function is measured with the Duke Activity Status Index (DASI). The DASI is a 12-item scale that measures physical function. Each question asks about whether the subject can complete a physical activity and are given the following options: Scores range from 0 to 58.2. Lower scores indicate lower levels of physical function.
Time Frame: Baseline, 24 weeks
Population: 92 participants in the Collaborative Care group were compared to 91 participants in the Usual Care group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
units on a scale | 8.96 [5.49 to 12.44] | 9.52 [6.10 to 12.94]
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = 5.59, 95% CI 2-sided [1.71 to 9.46]

9. Secondary Outcome: Change in Physical Health-related Quality of Life From Baseline to 24 Weeks
Description: Physical health-related quality of life is measured with the Short Form-12 Physical Component Score (SF-12 PCS). The SF-12 PCS a 6-item scale that assesses physical health-related quality of life. Each question provides the option of 2-6 answers. Some questions are Yes/No (2 options), while others ask how often something occurs (6 options, etc.). Scores are calculated using a formula and can range from 0 to 100. A score of 50 indicates average physical health-related quality of life. Higher scores represent higher than average physical health-related quality of life, and lower scores represent lower physical health-related quality of life.
Time Frame: Baseline, 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Collaborative Care | Usual Care
Number analyzed (Participants) | 92 | 91
units on a scale | 2.75 [0.20 to 5.31] | 4.21 [1.65 to 6.76]
Statistical Analysis 1: Comparison: Collaborative Care vs Usual Care; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis; Mean Difference (Final Values) = 2.30, 95% CI 2-sided [-0.54 to 5.14]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 24 weeks. Adverse events were inquired at each follow-up (6 weeks, 12 weeks, 18 weeks, 24 weeks).
Arm/Group | Collaborative Care | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/91
Other Adverse Events (participants affected / at risk) | 0/92 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No